CLINICAL TRIAL: NCT00608244
Title: A Phase II, Open-Label, Multi-Center Prospective, Conversion Study in Stable Liver Transplant Patients to Compare the Pharmacokinetics of LCP-Tacro Tablets Once-A-Day to Prograf® Capsules Twice-A-Day
Brief Title: Pharmacokinetics of LCP-Tacro in Stable Liver Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Veloxis Pharmaceuticals (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCP Tacro 2012
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2015-08-28 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Liver Failure
Keywords: Tacrolimus; Pharmacokinetics; Liver Transplantation
MeSH Terms: conditions — Liver Failure | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LCP-Tacro (Experimental): Prograf was administrated BID, doses per product labeling, with an interval of 12±1 hours between the morning and evening doses. Patients continued on the same dose from Day 0 through Day 7. On Day 8, all patients were converted to LCP Tacro QD for 14 Days with one fixed dose change allowed at Day 15. LCP-Tacro was administered orally once daily in the morning, with an interval of 24 ± 1 h between doses. Trough levels were to be maintained within predefined therapeutic ranges of 5 to 15 ng/mL.
  LCP-Tacro tablets were provided in 3 strengths: 1 mg, 2 mg, and 5 mg oral tablets.
  Interventions: Drug: LCP Tacro; Drug: Prograf

INTERVENTIONS:
Drug: LCP Tacro — In the morning of Day 8 (after completing one week treatment with Prograf), all patients will be converted to LCP Tacro QD with a conversion ratio of 0.66-0.8.
  LCP-Tacro will be administered for 14 Days with one fixed dose change allowed at Day 15. LCP-Tacro will be administered orally once daily in the morning, with an interval of 24 ± 1 h between doses.
  Trough levels were to be maintained within predefined therapeutic ranges of 5 to 15 ng/mL.
  Other Names: tacrolimus
Drug: Prograf — Prograf will be administrated twice a day, per product labeling, with an interval of 12 ± 1 hours between the morning and evening doses. Patients will continue on the same dose on Day 0 through Day 7 to maintain target trough levels of 5-12 ng/mL.
  Other Names: Tacrolimus

SUMMARY:
A three sequence, open-label, multi-center, prospective, study in stable liver transplant patients to assess and compare the pharmacokinetics (Cmax, C24, and AUC), and safety of LCP-Tacro (tacrolimus) tablets versus Prograf (tacrolimus) capsules.

DETAILED DESCRIPTION:
A three sequence, open-label, multi-center, prospective, study in stable liver transplant patients to assess and compare the pharmacokinetics (Cmax, C24, and AUC), and safety of LCP-Tacro (tacrolimus) tablets versus Prograf (tacrolimus) capsules.

Stable liver transplant patients who fulfill all I/E criteria will be enrolled and kept on Prograf for 7 days. Following a 24-hour PK study on Day 7 to determine pharmacokinetics for Prograf, all patients will be converted to once daily LCP-Tacro for 14 days with one fixed dose change allowed at Day 15.

On Day 14 and Day 21 a 24-hour LCP-Tacro PK study will be performed. On Day 22 patients will be converted back to their original twice daily dose of Prograf for a safety follow-up period of 30 days ending with a safety assessment on day 53.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years of age who are recipients of a liver transplant at least six months prior to enrollment
* Patients on oral Prograf therapy as part of their maintenance immunosuppression therapy, with stable doses and trough levels of tacrolimus of 5-12 ng/mL for at least four weeks prior to enrollment with at least two measurements at least two days apart in the screening period up to fourteen days prior to enrollment
* Concurrent immunosuppression with mycophenolate mofetil (MMF, CellCept) or mycophenolic acid delayed-release tablets (Myfortic) is allowed but patients on either of these medications should be on stable doses for at least four weeks prior to enrollment
* Patients with stable serum bilirubin, AST, ALT, and Alk Phos or GGT that are ≤ 2 times the upper limit of normal based on local laboratory criteria
* Patients with serum creatinine ≤2.0 mg/dL prior to enrollment
* Able to swallow study medication
* Patients capable of understanding the purposes and risks of the study, who can give written informed consent and who are willing to participate in and comply with the study protocol.
* Women of childbearing potential must have a negative serum pregnancy test within seven days prior to receiving study medication and agree to use contraceptive measures to avoid pregnancy during participation in the trial.

Exclusion Criteria:

* Recipients of any transplanted organ other than a liver
* White blood cell count ≤ 2.8 x 109/L
* Patients who are receiving a total dose of Prograf < 3 mg per 24 hours
* Patients who are receiving more than 10 mg of prednisone per day
* Patients unable or unwilling to provide informed consent
* Pregnant or nursing women
* Patients with reproductive potential who are unwilling/unable to use a double barrier method of contraception
* Administration of any other investigational agent in the three months prior to enrollment
* Patients receiving any drug interfering with tacrolimus metabolism
* Patients who have taken sirolimus within the three months prior to screening
* Patient with an episode of acute cellular requiring antibody therapy within the six months prior to enrollment
* Patients treated for acute cellular rejection within the thirty days prior to enrollment
* Patient who is HCV negative and has received an HCV positive (HCV RNA by PCR or HCV antibody) donor liver
* Patients presenting after liver transplantation with recurrent HCV infection, documented by presence of HCV RNA in serum and grade II or greater inflammation or stage II or greater fibrosis on liver biopsy
* Patients being actively treated with antiviral therapy, such as interferons or ribavirin, for recurrent hepatitis C.
* Patients with an alpha-feto protein ≥ 20 ng/mL
* Patient has a current malignancy or a history of malignancy (within the past five years), except basal or non-metastatic squamous cell carcinoma of the skin that has been treated successfully
* Patient has uncontrolled concomitant infection, a systemic infection requiring treatment, or any other unstable medical condition that could interfere with the study objectives
* Patient has severe diarrhea, vomiting, active peptic ulcer or gastrointestinal disorder that may affect the absorption of tacrolimus
* Patient will require therapy with any immunosuppressive agent other than those prescribed in the study
* Patient has a known hypersensitivity to corticosteroids or tacrolimus
* Patient has any form of current substance abuse (patients must pass a standard drug screen), psychiatric disorder or a condition that, in the opinion of the Investigator, may invalidate communication with the Investigator Version

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Alloway, PharmD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Alloway RR, Eckhoff DE, Washburn WK, Teperman LW. Conversion from twice daily tacrolimus capsules to once daily extended-release tacrolimus (LCP-Tacro): phase 2 trial of stable liver transplant recipients. Liver Transpl. 2014 May;20(5):564-75. doi: 10.1002/lt.23844. Epub 2014 Mar 26. PMID 24493215

RESULTS

PARTICIPANT FLOW:
Groups:
- LCP-Tacro: All Patients received Prograf for 7 days, then all patients were converted to once daily LCP-Tacro for 14 days. One dose adjustment up or down 25% was permitted on Day 15.
  On Day 22, patients were converted back to their original twice daily dose of Prograf for a safety follow-up period of 30 days.
  LCP-Tacro 1 mg, 2 mg and 5 mg tablets administered orally QD, dosing per conversion algorithm to maintain tacrolimus trough concentrations between 5 to 15 ng/mL.
Period: Overall Study
Arm/Group | LCP-Tacro
Started | 59
Completed | 57
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Low trough levels | 1

BASELINE CHARACTERISTICS:
Groups:
- LCP-Tacro: Evaluation of steady state tacrolimus exposure (AUC0-24) and trough levels (C24) in stable liver transplant recipients converted from Prograf to LCP-Tacro in a 3-sequence study design and validate the dose conversion ratio determined in the Phase 1 program.
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (11.15)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 59
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 8
  White | 46
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Steady State Tacrolimus Trough Levels (C24).
Description: Patients had a baseline trough level (C24) measured at day 7 before conversion to LCP-Tacro.
Time Frame: 7 Days
Population: The arithmetic mean and standard deviation is given.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Prograf: Prograf 0.5 mg, 1 mg and 5 mg capsules administered orally twice daily, dosing per conversion algorithm to maintain tacrolimus trough concentrations between 5 to 15 ng/mL.
Arm/Group | Prograf
Number analyzed (Participants) | 57
ng/mL | 6.72 (2.07)

2. Primary Outcome: Evaluation of Steady State Tacrolimus Exposure (AUC 0-24).
Description: Patients had a baseline AUC measured (0 to 24 hours) at day 7 before conversion to LCP-Tacro.
  The following time points were used to obtain the PK curve for Prograf on day 7: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 12.5, 13, 13.5, 14, 15, 16, 20 and 24 hours after the morning dose.
Time Frame: 7 Days
Population: The arithmetic mean and standard deviation is given.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Prograf
Number analyzed (Participants) | 57
ng*hr/mL | 205.14 (61.0)

3. Primary Outcome: Evaluation of Steady State Tacrolimus Exposure Trough Levels (C24).
Description: Patients were converted from Prograf to LCP-Tacro on day 7. On day 21, a trough level (C24) was measured.
Time Frame: 21 Days
Population: 57 completed the study but one patient was excluded from the PP analysis due to low trough levels.
  The arithmetic mean and standard deviation is given.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- LCP-Tacro: LCP-Tacro 1 mg, 2 mg and 5 mg tablets administered orally QD, dosing per conversion algorithm to maintain tacrolimus trough concentrations between 5 to 15 ng/mL.
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 56
ng/mL | 6.85 (2.63)

4. Primary Outcome: Evaluation of Steady State Tacrolimus Exposure (AUC 0-24) on Day 21.
Description: Patients were converted from Prograf to LCP-Tacro on day 7. On day 21, AUC was measured (0 to 24 hours).
  The following time points were used to obtain the PK curve for LCP-Tacro on day 21: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20 and 24 hours post-dose.
Time Frame: 21 Days
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 56
ng*hr/mL | 215.66 (79.40)

5. Primary Outcome: Safety Evaluation
Description: A combination of deaths, graft failure and biopsy proven acute rejections (BPAR) was used to evaluate the safety.
Time Frame: 52 days
Population: All enrolled patients are included in the safety population.
Measure: Number; unit: participants
Arm/Group | LCP-Tacro
Number analyzed (Participants) | 59
participants
  Death | 0
  Graft Failure | 0
  BPAR | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of first dose of study drug and until the end of the follow up period at day 52.
Groups:
- LCP-Tacro: LCP-Tacro 1 mg, 2 mg and 5 mg tablets administered orally QD, dosing per conversion algorithm to maintain tacrolimus trough concentrations between 5 to 15 ng/mL.
  59 patients were enrolled into the study and all 59 were dosed with LCP-Tacro.
- Prograf: Prograf 0.5 mg, 1 mg and 5 mg capsules administered orally twice daily, dosing per conversion algorithm to maintain tacrolimus trough concentrations between 5 to 15 ng/mL.
  59 patients were enrolled into the study and all 59 were dosed with Prograf. Adverse Events occurring during the follow up period (Days 22-51) have been counted in the Prograf treatment arm as patients were on Prograf during this period.
Arm/Group | LCP-Tacro | Prograf
Serious Adverse Events (participants affected / at risk) | 1/59 | 0/59
Other Adverse Events (participants affected / at risk) | 19/59 | 7/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=59) | Prograf (N=59)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LCP-Tacro (N=59) | Prograf (N=59)
Fatigue (General disorders) | 6 (8) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (3) | 2 (2)
Contusion (Investigations) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Tremor (Nervous system disorders) | 3 (3) | 1 (1)
Liver function test abnormal (Investigations) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This study is a multicenter collaborative investigation and the clinical trial results are to be published as a collaborative manuscript. Authorship will reflect varying levels of individual contribution to the study by the individual PIs.